CLINICAL TRIAL: NCT03062150
Title: Effects of Mineralocorticoid Receptor Stimulation on Cognitive Bias and Social Cognition in Patients With Major Depression and Healthy Controls: What's the Role of NMDA Receptors?
Brief Title: Mineralocorticoid Receptor, NMDA Receptor and Cognitive Function in Depression
Acronym: MISO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Prof. Dr. Christian Otte, Professor of Psychiatry, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: OT 209/7-1; 2014-005239-15 (EudraCT Number)
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fludrocortisone; Cycloserine

STUDY DESIGN:
Intervention Model Description: randomized double-blind placebo-controlled parallel group design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo+Placebo (Placebo Comparator): Placebo: pill, 8mm, single dose, Lichtenstein, Winthrop Arzneimittel GmbH.
  Interventions: Drug: Placebo
- Fludrocortisone+Placebo (Active Comparator): Fludrocortisone: pill, Astonin H 0,1gm, single dose, Merck Serono GmbH
  Placebo: pill, 8mm, single dose, Lichtenstein, Winthrop Arzneimittel GmbH.
  Interventions: Drug: Placebo; Drug: Fludrocortisone
- Placebo+D-Cycloserine (Active Comparator): Placebo: pill, 8mm, single dose, Lichtenstein, Winthrop Arzneimittel GmbH.
  D-Cycloserine: capsule, Cycloserine 250mg, single dose, King Pharmaceuticals Ltd
  Interventions: Drug: Placebo; Drug: D-Cycloserine
- Fludrocortison+D-Cycloserine (Active Comparator): Fludrocortisone: pill, Astonin H 0,1gm, single dose, Merck Serono GmbH
  D-Cycloserine: capsule, Cycloserine 250mg, single dose, King Pharmaceuticals Ltd
  Interventions: Drug: Fludrocortisone; Drug: D-Cycloserine

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Fludrocortisone+Placebo; Placebo+D-Cycloserine; Placebo+Placebo
Drug: Fludrocortisone — Fludrocortisone
  Arms: Fludrocortison+D-Cycloserine; Fludrocortisone+Placebo
Drug: D-Cycloserine — D-Cycloserine
  Arms: Fludrocortison+D-Cycloserine; Placebo+D-Cycloserine

SUMMARY:
The steroid hormone cortisol is released in response to stress and acts in the central nervous system upon glucocorticoid (GR) and mineralocorticoid receptors (MR). GR are widely distributed across the brain while MR are predominantly expressed in the hippocampus and prefrontal cortex - two brain areas closely related to memory and executive function. Stimulation of MR leads to an increase of glutamate that act on glutamatergic NMDA receptors in the hippocampus and prefrontal cortex. In previous studies, the investigators have shown that fludrocortisone, a mineralocorticoid receptor (MR) agonist, improves memory and executive function in depressed patients and healthy controls. However, depressed patients not only exhibit cognitive deficits in traditional neuropsychological domains such as memory or executive function. In addition, there are depression-specific alterations such as cognitive bias and deficits in social cognition, two clinically highly relevant areas. Therefore, the specific aims of this renewal proposal are two-fold:

* To examine whether beneficial effects of fludrocortisone in depressed patients can be extended to depression-specific cognitive bias and to social cognition
* To determine whether beneficial effects of fludrocortisone depend on NMDA-receptor function and whether these beneficial effects can be enhanced by NMDA receptor stimulation.

The investigators hypothesize that fludrocortisone will improve cognitive bias and social cognition in depressed patients and that its beneficial effects depend on the NMDA receptor. Therefore, the investigators further hypothesize that the effects of fludrocortisone can be enhanced by co-administration of the partial NMDA receptor agonist D-cycloserine.

The study not only advances current knowledge by further examining the mechanism of action by which MR stimulation exerts beneficial effects on cognition but extends these effects to depression-specific cognitive bias and alterations in social cognition. Furthermore, a potential interaction between MR and NMDA receptors is highly clinically relevant given the promising results with NMDA receptor antagonists in the treatment of major depression.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Depressed male and female patients according to DSM-V & minimum of 17-items Hamilton Depression Score of 18
* healthy controls
* informed consent signed

Exclusion Criteria:

* Current use of antidepressants, antipsychotics, or mood stabilizer
* Relevant medical or neurological disorders
* Pregnancy or unsure contraception
* Relevant psychiatric comorbidity (bipolar or psychotic disorders)
* Active alcohol or other substance abuse/dependance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Emotional dot probe | 1 hour
  In this task, two stimuli (each a photography of a face) are presented quickly on a computer screen (500 ms), and one face stimulus is replaced by a probe (1100 ms). Face pictures can show a sad, happy or neutral expression and are paired as neutralneutral, neutral-sad, or neutral-happy. Participants respond as fast as possible by pressing a key to correspond to the location of the probe.
  Attentional bias can be derived by the average reaction time when the probe replaces negative stimuli (sad faces), the average reaction time when the probe replaces neutral stimuli (neutral faces), and the average reaction time of positive (happy faces) and neutral stimuli (neutral faces).

SECONDARY OUTCOMES:
Facial recognition task | 1 hour
  This emotion recognition task features two basic emotions - sadness and anger - and a number of control trials containing neutral face expressions. Overall, 6 male and 6 female faces were taken from the NIMSTIM scale (Tottenham et al. (2009); http://www.macbrain.org/resources.htm).
  Two graduations from the full emotion (100%) were created (40% and 80%) and are presented in 24 trials per percentile rank in shades of grey. In addition, 24 control Trials are presented with 0% (neutral) emotion. Overall, the task contains 120 trials in randomized order. Each face is shown for 1 second and is replaced by a grey screen, which requests an answer by showing the three possible answers (sadness, anger, neutral). This screen is presented for 4 seconds and participants make their Responses by pressing one of three keys on the keyboard (arrow keys). Reaction time and correct responses are measured.
Multifaceted Empathy Test (MET) | 1 hour
  To assess cognitive and emotional empathy, the MET will be used (Dziobek et al , 2008) in a modified version (Hurlemann et al , 2007; Dziobek et al , 2011; Ritter et al , 2011). The MET is a PC-assisted test consisting of photographs that show 30 picture Stimuli with people in emotionally charged situations. To assess cognitive empathy, participants will be required to infer the mental state of the subject in the photo and will be asked to indicate the correct one from a list of four. To assess emotional empathy, participants will be asked to rate the degree of empathic concern they feel for the person in the Picture (Likert scale, 1 = not at all, 9 = very much).
Virtual Water Maze | 1 hour
  Participants are placed in a virtual reality, presented on a computer screen, consisting of a room with a pool in the center. In the pool, there is an invisible platform, that participants have to reach as fast as possible. Participants can move in an ego-perspective with a joystick. In several trials, participants learn to reach the platform. The better participants learn, the faster they reach the platform and the shorter is the path they used.
  In the last trial, participants do not get to know whether they reached the platform. The time (sec) spent in the right quadrant, is the outcome measurement, used to determine visuospatial memory.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Otte, MD, Principal Investigator — Charité University Medical Center Berlin, Dept. of Psychiatry
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Otte C, Wingenfeld K, Kuehl LK, Kaczmarczyk M, Richter S, Quante A, Regen F, Bajbouj M, Zimmermann-Viehoff F, Wiedemann K, Hinkelmann K. Mineralocorticoid receptor stimulation improves cognitive function and decreases cortisol secretion in depressed patients and healthy individuals. Neuropsychopharmacology. 2015 Jan;40(2):386-93. doi: 10.1038/npp.2014.181. Epub 2014 Jul 18. PMID 25035081
- [Background] Hinkelmann K, Wingenfeld K, Kuehl LK, Fleischer J, Heuser I, Wiedemann K, Otte C. Stimulation of the mineralocorticoid receptor improves memory in young and elderly healthy individuals. Neurobiol Aging. 2015 Feb;36(2):919-24. doi: 10.1016/j.neurobiolaging.2014.09.008. Epub 2014 Sep 16. PMID 25442112
- [Background] Otte C, Wingenfeld K, Kuehl LK, Richter S, Regen F, Piber D, Hinkelmann K. Cognitive function in older adults with major depression: Effects of mineralocorticoid receptor stimulation. J Psychiatr Res. 2015 Oct;69:120-5. doi: 10.1016/j.jpsychires.2015.08.001. Epub 2015 Aug 4. PMID 26343603
- [Derived] Nowacki J, Wingenfeld K, Kaczmarczyk M, Chae WR, Abu-Tir I, Deuter CE, Piber D, Hellmann-Regen J, Otte C. Cognitive and emotional empathy after stimulation of brain mineralocorticoid and NMDA receptors in patients with major depression and healthy controls. Neuropsychopharmacology. 2020 Dec;45(13):2155-2161. doi: 10.1038/s41386-020-0777-x. Epub 2020 Jul 28. PMID 32722659